CLINICAL TRIAL: NCT01209910
Title: Effects of Free Water Protocol on Inpatients in a Neurological Rehabilitation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. S. Pooyani, Assistant professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0120
Record Dates: First submitted 2010-07-13; First posted 2010-09-27 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Water; Drinking Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- free water (Experimental): The subjects in this arm will be able to drink water followings study rules.
  Interventions: Other: Water
- Control (No Intervention): These subjects will be observed during the study.

INTERVENTIONS:
Other: Water — Subjects in this arm will be able to drink water with some conditions.
  Other Names: Drinking water
  Arms: free water

SUMMARY:
Inpatients in the neurology rehabilitation units at Riverview Health Center- people who are brain-injured and or who have had a stroke - often have dysphagia as a result of their condition. They are considered at high risk of aspiration, which can result in pneumonia. To limit that risk, these patients are only allowed to consume thickened liquids at the beginning of their rehabilitation. They are restricted from consuming thin liquids, which means they can't even drink water. Depending on the rate of their rehabilitation, these restrictions can last from six months to a year.

Patients on a diet of thickened liquids sometimes have difficulty consuming the required daily intake of fluids and they become dehydrated, which in turn can lead to other health complications. As well, thickened liquids do not always satisfy a patient's thirst, says Pooyania.

While Riverview does not allow inpatients with dyspagia to have water at the beginning of their rehabilitation, many rehab facilities in Canada and the U.S. follow the "Frazier Free Water Protocol," which does allow patients unrestricted water intake prior to and 30 minutes after meals. The belief that this protocol is safe is based on research done at the Frazier Rehabilitation Institute, where a study demonstrated no difference in rates of aspiration pneumonia between an experimental group on a free water protocol and a control group.

The Frazer study was only one randomized controlled trial with a very limited number of patients. There have been a few case reports as well, but at Riverview centre, the protocol is not accepted because the investigators don't believe there is enough evidence behind it. The investigators intend to provide more clinical evidence so that both the risks and benefits of a free water protocol can be assessed.

The investigators will be screening patients admitted to the neurology rehabilitation units at RCH, including both the stroke and acquired brain injury programs. The investigators expect to find at least 30 suitable candidates.

Participants will be educated about dysphagia and the free water protocol, and the treatment group will be allowed unrestricted water intake prior to and 30 minutes after meals. Individualized intervention to minimize aspiration will be provided. Daily and weekly monitoring and testing of all patients will take place. The pilot study will continue for 11 months. A secondary objective of the research is to determine the feasibility of expanding into a multi-centre clinical trial

DETAILED DESCRIPTION:
Research to determine the impact of a free water protocol on inpatients in a neurological rehabilitation setting is extremely relevant to the patient population at Riverview Health Centre (RHC), as many patients at RHC receive a modified diet consisting of thickened liquids. To date, the research base for the use of free water protocols is limited. Despite the general lack of research evidence, modified versions of a free water protocol have been adopted at numerous facilities across North America. Pursuing clinical research to measure the effects of a free water protocol on rate of aspiration pneumonia, quality of life related to swallowing, fluid intake, and hydration levels, would provide research evidence to help guide patient care. If such research were to show that a free water protocol could be used without increased risk to patients with dysphagia, the patient population at Riverview, and at other rehabilitation centers, could benefit.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with thin fluid restriction to the Stroke and Acquired Brain Injury Units at Riverview Health Centre for the duration of the study will be considered for eligibility.

Exclusion Criteria:

* Exclusion criteria include the following: history of severe pulmonary complications, individuals demonstrating severe coughing to the point of discomfort or medical complications when consuming thin fluids, individuals with immune deficiency problems or severe cognitive impairment that would affect patient's ability to sign the consent form or follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Outcome measures will include the rate of aspiration pneumonia, quality of life related to swallowing, fluid intake, and hydration level | While admitted in hospital, or develop a complication up to 12 months
  Outcome measures will include the rate of aspiration pneumonia, quality of life related to swallowing, fluid intake, and hydration level

SECONDARY OUTCOMES:
to expand the study to a multi-centre clinical trial. | one year
  to expand the study to a multi-centre clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Pooyania, MD. FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada